CLINICAL TRIAL: NCT06183463
Title: Use of Reconstructive Surgery for Women Consulting in Sexology at the University Hospitals of Strasbourg for Sexual Mutilation
Brief Title: The Use of Reconstructive Surgery for Sexually Mutilated Women at the University Hospitals of Strasbourg
Acronym: Repair-SM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8724
Record Dates: First submitted 2023-12-13; First posted 2023-12-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Sexual Trauma
Keywords: Sexual mutilation
MeSH Terms: conditions — Sexual Trauma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Despite awareness since the 1980s and a legal framework to punish sexual mutilation, this tradition continues in many countries, particularly in Africa but not only in the Middle East, Malaysia and Indonesia. This custom, carried out among increasingly young little girls, exposes them to infectious, hemorrhagic and even death risks and sometimes significant obstetric complications.

Every year, 3 million girls and young women are sexually mutilated around the world, or one woman every 15 seconds.

In recent years, a surgical repair technique has been created by a French urologist, Professor Foldès. This technique allows clitoral reconstruction. Sensory reacquisition after this intervention may take a few months, but the functional results are quite good.

There is little or no data concerning the use of reconstructive surgery for these mutilated patients consulting in sexology and the future of patients post-operatively or who have not had recourse to reconstructive surgery. The investigators then questioned the decision of these patients and their future.

ELIGIBILITY:
Inclusion Criteria:

* Adult woman (≥18 years old)
* having consulted sexology at the HUS for sexual mutilation between 01/01/2011 and 12/31/2021.
* having had clitoral repair surgery at the HUS between 01/01/2011 and 12/31/2021
* not objecting, after information, to the reuse of their data for the purposes of this research

Exclusion Criteria:

* Woman who expressed her opposition to participating in the study
* impossibility of providing the subject with informed information (difficulties in understanding the subject, etc.)
* Woman under judicial protection or under guardianship or curatorship.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult woman (≥18 years old) having consulted sexology at the HUS for sexual mutilation between 01/01/2011 and 12/31/2021.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Estimated)
Dates: Start 2022-11-24 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the future of patients who consulted sexology for sexual mutilation between 2011 and 2021 at the HUS, whether or not they opted for reconstructive surgery. | Through study completion, an average of 6 months
  This assessment is made via a questionnaire of nine questions relating to their future.

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Assistance Médicale à la Procréation - CHU de Strasbourg - France, Strasbourg, France